CLINICAL TRIAL: NCT05084677
Title: Toripalimab Combined With Concurrent Platinum-based Chemoradiotherapy in Patients With Locally Advanced Cervical Cancer: An Open-Label, Single-Arm, Phase II Trial
Brief Title: Toripalimab Combined With Concurrent Chemoradiotherapy in Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202020080608084322319
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 arm (Experimental): PD-1 concurrent with and subsequent after concurrent chemoradiotherapy
  Interventions: Combination Product: Toripalimab Combined With Concurrent Platinum-based Chemoradiotherapy

INTERVENTIONS:
Combination Product: Toripalimab Combined With Concurrent Platinum-based Chemoradiotherapy — Toripalimab 240mg intravenously(IV) every 3 weeks (Q3W) concurrent with chemoradiotherapy; 6 cycles of Toripalimab 240mg intravenously(IV) every 3 weeks (Q3W) after chemoradiotherapy; Toripalimab 240mg intravenously(IV) every 6 weeks (Q6W) thereafter until the whole treatment period reached one year since the beginning.

SUMMARY:
To explore the efficacy and tolerance of adding toripalimab simultaneously and subsequently to concurrent platinum-based chemoradiotherapy in patients with locally advanced cervical cancer.

DETAILED DESCRIPTION:
Up to now, there have been several prospective studies exploring the effectiveness of PD-1 inhibitors in patients with recurrent/ metastatic cervical cancer. The results showed that the overall objective response rate (ORR) was between 12.2% and 55.6%, and pembrolizumab was approved by the US Food and Drug Administration for patients with advanced PD-L1-positive cervical cancer who experienced progression during or after chemotherapy. However, the evidence of using PD-1 inhibitors together with concurrent chemotheradiotherapy in patients with locally advanced cervical cancer is rare, so we initiated this single arm prospective phase II clinical study. The purpose is to explore the efficacy and tolerance of adding toripalimab simultaneously and subsequently to concurrent chemoradiotherapy in patients with locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75;
* Untreated patients with pathologically proven locally advanced cervical cancer;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Adequate hematological, renal and hepatic functions:

  1. Hemoglobin > 8.0 g/dl
  2. Neutrophils > 2000 cells/μl; Leukocytes > 4 × 109/L
  3. Platelets > 100 × 109/L

  g. Serum urea nitrogen (BUN) ≤ 1.5 × upper normal limit (UNL) h. Serum creatinine (Cr) ≤ 1.5 × upper normal limit (UNL) d. Serum ALT/AST ≤ 2.5× UNL e. Serum Total bilirubin ≤ 1.5× UNL
* Life expectancy > 6 months
* Eligible for concurrent chemoradiotherapy assessed by principle investigator;
* No obvious active bleeding;
* Written informed consent must be available before study registration

Exclusion Criteria:

* Recurrent or distant metastatic disease;
* Prior malignancies (other than curable non-melanoma skin cancer) within 5 years;
* Active autoimmune diseases requiring systemic treatment or other diseases requiring long-term use of substantial amount of hormones or other immunosuppressants;
* Patients who need to receive systemic corticosteroids (dose equivalent to or higher than prednisone 10mg qd) or other immunosuppressants within 14 days before enrollment or during the study;
* Vaccination of live attenuated vaccine 30 days before enrollment, or planned vaccination of live attenuated vaccine during the study;
* Previous organ transplantation or HIV patients;
* Allergic to macromolecular proteins /monoclonal antibodies, or to any test drug component;
* Active acute or chronic viral hepatitis B or C. Hepatitis B virus (HBV) DNA> 2000IU/ml or 104 copies/ml; hepatitis C virus (HCV) RNA> 103 copies/ml.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 1 year
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) using RECIST v1.1

SECONDARY OUTCOMES:
Progression free survival | 2 years
  Time from diagnosis of disease to disease progression or death due to any cause
Overall survival | 3 years
  Time from diagnosis of disease of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute&Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Li C, Cao Y, Zhu L, Zhang B, You J, Hou H, Wang J, Yuan Z. Toripalimab combined with concurrent platinum-based Chemoradiotherapy in patients with locally advanced cervical Cancer: an open-label, single-arm, phase II trial. BMC Cancer. 2022 Jul 19;22(1):793. doi: 10.1186/s12885-022-09866-w. PMID 35854236